CLINICAL TRIAL: NCT06800118
Title: The Effect of Music on Anxiety and Vasospasm in Patients Undergoing Transradial Angiography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Nida Aykuş Yeşil, Graduate Nursing Student, Mersin University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MersinU-HEM-NY-01
Record Dates: First submitted 2025-01-19; First posted 2025-01-29 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Radial Artery Spasm; Anxiety; Music Therapy
Keywords: Radial artery spasm; anxiety; music therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Music will be played for the patients in this group during transradial coronary angiography.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Active Comparator): In addition to standard care, patients in the intervention group will listen to music through headphones at a volume adjusted to their preference. The selected music will feature Classical Turkish Music performed on the ney in the Hüseyni maqam, which has been shown in previous studies to promote relaxation.
  Interventions: Device: Music intervention
- control group (No Intervention): Patients in the control group will receive standard care, including obtaining informed consent, recording medical history, establishing venous access, measuring vital signs, and performing an ECG. After the procedure, the wrist sheath will be removed, bleeding control will be performed, and the wrist will be dressed with a pressure bandage. Patients without percutaneous coronary intervention will be discharged 6 hours post-procedure, while those with percutaneous coronary intervention will remain under observation for one day.

INTERVENTIONS:
Device: Music intervention — Music will be played for patients undergoing coronary angiography, and vasospasm and pain levels will be evaluated.
  Arms: intervention group

SUMMARY:
Cardiovascular diseases are among the most significant health issues threatening human well-being, representing the leading cause of mortality and morbidity worldwide and in our country among non-communicable diseases. In Turkey, 33.4% of deaths are attributed to circulatory system diseases and ischemic heart diseases, with coronary artery disease (CAD) being the most common cause. The most frequently applied and accurate invasive diagnostic method for diagnosing CAD is coronary angiography.

Coronary angiography, still regarded as the gold standard today, is a diagnostic procedure that visualizes the heart's blood vessels using contrast media. This procedure can be performed via the femoral, brachial, radial, or axillary arteries. In the past, coronary interventional procedures were commonly performed through the femoral artery. However, following the 2017 European Society of Cardiology (ESC) guidelines on ST-segment elevation myocardial infarction (STEMI) management, the radial artery has become the preferred route due to its lower risk of bleeding and shorter hospital stays. Coronary angiography is performed in a sterile environment while the patient is awake.

Due to its invasive nature and the involvement of a vital organ, coronary angiography can evoke anxiety and fear of death in patients. Factors contributing to this include uncertainty about the procedure, unfamiliarity with the environment, communication with unknown personnel, exposure to medical terminology, and unusual sounds in the procedure room.

The radial artery is more prone to vasospasm than other vessels used in coronary angiography, due to its smaller diameter and rich smooth muscle content. Local anesthesia is administered at the access site to reduce pain during radial artery interventions. Additionally, anticoagulant and vasodilatory drugs are used to prevent procedure-related vasospasms and thrombotic events. Despite these preventive measures, vasospasm is observed in 4-20% of patients undergoing transradial coronary angiography.

Anxiety experienced by patients during the procedure can also contribute to vasospasm in the radial artery. Various invasive and non-invasive interventions, such as listening to music, acupressure, and massage, are frequently employed to reduce patient anxiety. Among these non-invasive methods, providing music during the procedure has gained prominence. Music helps divert patients' attention, enabling them to distance themselves from pain, fear, stress, and anxiety.

DETAILED DESCRIPTION:
Type of Study This study is designed as a prospective, two-arm (1:1), randomized controlled clinical trial. The randomized controlled trial will be reported in accordance with the CONSORT guidelines.

Study Setting and Characteristics The study will be conducted in the Coronary Angiography Unit of Mersin University Faculty of Medicine Hospital's Cardiology Clinic. The Coronary Angiography Unit is equipped with eight day-patient beds and two angiography devices. Eight nurses work in this unit between 08:00 and 16:00. Patients scheduled for coronary angiography are admitted to the hospital on the morning of the procedure.

Patients visit the Cardiology outpatient clinic to schedule their coronary angiography, and preparations are carried out in the Coronary Angiography Unit upon their arrival on the day of the procedure. These preparations include obtaining the patient's medical history and informed consent, establishing venous access, measuring vital signs, and performing an electrocardiogram (ECG), which is added to the patient's file. Before the procedure, oral intake is restricted for 4 hours. After the procedure, the arterial sheath in the wrist is removed by the physician immediately after the patient is transferred to their bed. Hemostasis is achieved, and the wrist is covered with a pressure bandage.

If no percutaneous coronary intervention is performed, bleeding control is assessed 6 hours post-procedure, and the patient is discharged. If a percutaneous coronary intervention is performed, the patient is monitored in the cardiology clinic for one day post-procedure.

Randomization and Blinding A total of 90 patients, meeting the inclusion criteria, will be randomized into two groups (A and B) using a computer-generated randomization table prepared by a statistician. The designation of group A or B as the intervention or control group will be determined by a coin toss at the beginning of the study. Information regarding patient group assignments, based on the randomization table, will be placed in opaque envelopes and securely stored by the advisor. Upon initiating the procedure, the investigator will open the envelope after obtaining the patient's informed consent to determine the group assignment. The investigator will be blinded to group assignments, but patients and the investigator cannot be blinded due to the nature of the intervention (music listening). Data will be recorded in a blinded manner, and analysis will be performed by an independent statistician who is unaware of group assignments.

Expected Outcomes and Data Collection Forms The primary outcome of the study is to evaluate the effect of music on anxiety in patients undergoing transradial coronary angiography. The secondary outcome is to assess the effect of music on radial vasospasm.

Data will be collected using the following forms:

Demographic Information Form: This form includes patient demographic characteristics such as age, sex, marital status, educational level, and presence of chronic diseases.

State Anxiety Inventory (STAI): This validated inventory, originally developed by Spielberger et al. and adapted into Turkish by Öner and Le Comte, measures anxiety levels. The STAI includes 20 items assessing how individuals feel at a specific moment, with scores ranging from 20 to 80. Higher scores indicate greater anxiety. Scores are categorized as follows: 0-19 (no anxiety), 20-39 (mild anxiety), 40-59 (moderate anxiety), and 60-79 (severe anxiety). Scores above 60 suggest a need for professional support.

Radial Vasospasm Evaluation Form: This form includes information on the reason for coronary angiography, the occurrence of radial vasospasm during the procedure, and its associated symptoms.

Data Collection Process After obtaining ethical approval, data will be collected between October 1, 2024, and April 1, 2025. Patients meeting the inclusion criteria will complete the informed consent form, the Demographic Information Form, and the STAI before the procedure. The Coronary Angiography Unit will designate one room for the music intervention group and another for the control group.

Control Group: Patients in the control group will receive standard care, including obtaining informed consent, recording medical history, establishing venous access, measuring vital signs, and performing an ECG. After the procedure, the wrist sheath will be removed, bleeding control will be performed, and the wrist will be dressed with a pressure bandage. Patients without percutaneous coronary intervention will be discharged 6 hours post-procedure, while those with percutaneous coronary intervention will remain under observation for one day.

Intervention Group: In addition to standard care, patients in the intervention group will listen to music through headphones at a volume adjusted to their preference. The selected music will feature Classical Turkish Music performed on the ney in the Hüseyni maqam, which has been shown in previous studies to promote relaxation.

All patients will complete the STAI again immediately after the procedure. The same physician will perform all coronary angiography procedures using the same equipment and catheters. Radial artery vasospasm will be identified by symptoms such as progressive forearm pain, increased pain during catheter manipulation, resistance during catheter manipulation, and sheath movement-related resistance and pain. At least two of these symptoms must be present to confirm radial artery vasospasm. Information regarding vasospasm occurrence will be obtained from the physician and recorded on the Radial Vasospasm Evaluation Form.

Music listening, a non-invasive and independent nursing intervention, will be terminated immediately if any adverse effects are observed.

Data Analysis Data will be analyzed using appropriate statistical methods. Descriptive statistics will include frequency, percentage, mean, and standard deviation. Parametric or non-parametric tests will be used to compare data based on normality distribution.

Ethical Considerations Prior to the study, written ethical approval will be obtained from the Clinical Research Ethics Committee of Mersin University and the Department of Cardiology at Mersin University. Written informed consent will be obtained from all participants. The study will be conducted in accordance with the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Indication for radial coronary angiography (CA) due to non-acute coronary syndrome (ACS) reasons
* Undergoing coronary angiography for the first time
* Aged 18 years or older
* Conscious, oriented, and cooperative
* Able to read and understand Turkish
* Willing to participate in the study
* Without any physical limitations preventing music listening
* Without a diagnosis of hearing loss
* Not using a hearing aid
* Without a diagnosis of anxiety disorder
* Without any mental health disorders
* Having signed the "Voluntary Informed Consent Form.

Exclusion Criteria:

* Indication for radial coronary angiography (CA) due to acute coronary syndrome (ACS)
* Previous history of coronary angiography
* Under the age of 18,
* Unconscious, disoriented, or uncooperative,
* Unable to read or understand Turkish,
* Unwilling to participate in the study,
* Having physical limitations that prevent listening to music,
* Diagnosed with hearing loss,
* Using a hearing aid,
* Diagnosed with an anxiety disorder or taking medication for anxiety,
* Having a mental health disorder,
* Not signing the "Voluntary Informed Consent Form."

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
the State-Trait Anxiety Inventory (STAI) | day 1
  The STAI (State-Trait Anxiety Inventory) is a psychological tool developed to assess individuals' anxiety levels and consists of a total of 40 questions. The scale addresses anxiety in two distinct dimensions: State Anxiety and Trait Anxiety. State anxiety measures the individual's temporary level of anxiety in response to a specific and transient situation, while trait anxiety evaluates the individual's general tendency to experience anxiety and their predisposition to perceive anxiety as a personality trait. Both subscales consist of 20 questions, and individuals are asked to indicate how much the given statements apply to them.

CONTACTS AND LOCATIONS:
Overall Officials: Nida YESİL, Graduate Nursing Student, Principal Investigator — Mersin University Faculty of Nursing
Locations (1):
- Mersin Universiy Faculty of Nursing, Mersin, yenisehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided